CLINICAL TRIAL: NCT04560803
Title: Using Autologous Epidermal Skin Micrografts to Improve Healing In Radiation Wounds: A Pilot Study
Brief Title: Epidermal Skin Grafts to Improve Healing In Radiation Wounds
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Collaborators: 3M (Industry)
Responsible Party: Principal Investigator, Thanh-Nga T. Tran, M.D.,Ph.D., Instructor, Massachusetts General Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2019P001728
Record Dates: First submitted 2020-09-17; First posted 2020-09-23 (Actual); Last update posted 2023-10-23 (Actual); Status verified 2023-10

CONDITIONS: Radiation Dermatitis
Keywords: Epidermal graft; Skin graft; Radiation wound
MeSH Terms: conditions — Radiodermatitis

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Epidermal Grafting (Experimental): This irradiated area of the skin will be treated with autologous epidermal grafts
  Interventions: Device: CelluTomeTM Epidermal Harvesting System
- No treatment (No Intervention): This irradiated area will not receive any treatment

INTERVENTIONS:
Device: CelluTomeTM Epidermal Harvesting System — Autologous epidermal grafts that will be placed at the treatment site
  Arms: Epidermal Grafting

SUMMARY:
Patients undergoing radiation for the treatment of malignancies may suffer from side effects to the skin in the form of radiation dermatitis. This can lead to local wound formation with poor healing. Treatment options for the resulting wound can range from watchful waiting to more aggressive debridement and secondary grafting.

Epidermal grafting is a technique in which autologous epidermis is used to cover wounds that are larger than the donor site. Previous studies have demonstrated that this is an effective treatment for different wounds and ulcers but its utility has not yet been evaluated for the treatment of radiation induced injuries.

The CelluTome Epidermal Grafting System is a semi automated device that allows easy formation of epidermal Blister.

Our study will evaluate the efficacy of epidermal grafts collected using the CelluTome device in the treatment of radiation dermatitis.

DETAILED DESCRIPTION:
Patients participating in this study will undergo the epidermal grafting procedure to a part of their radiation-induced wound. The remaining untreated area will serve as an irradiated control.

The donor tissue will be collected from normal skin in the upper thigh area. In addition to their primary screening visit, patients will be followed up closely in a series of 9 study visits. During these sessions, photographs will be taken and patients will be asked to fill out questionnaires.

ELIGIBILITY:
Inclusion Criteria:

* Status post radiation treatment, with radiation-induced wound. This includes patient with moist desquamation as well as full epidermal necrosis and superficial dermal ulcerations, this wound would otherwise be allowed to heal by secondary intention;
* Having suitable areas of treatment: All wounds in the area of interest must be at least 20 cm2 (~10 cm2 per treatment/control area);
* The radiation injury must have a suitable adjacent irradiated control site before initiation of treatment. This will be determined by objective measurements of % wound epithelization, wound erythema, pliability, induration and thickness at enrollment;
* Able and willing to comply with all visit, treatment and evaluation schedules and requirements;
* Wound considered appropriate by physician to receive epidermal grafting;
* Able to understand and provide written informed consent;

Exclusion Criteria:

* Active tanning, including the use of tanning booths, during the course of the study;
* Study wound exhibits clinical signs and symptoms of infection at the screening/enrollment visit;
* Patient unable to provide donor site for epidermal harvesting;
* Wound sites located on the face, hands or feet
* Adverse reactions to compounds of any external agent (e.g., gels, lotions or anesthetic creams) required for use in the study, if no alternative to the said agent exists;
* History of collagen vascular disease;
* Active Herpes Simplex or Zoster at the time of treatment or having experienced more than three episodes of Herpes Simplex / Zoster eruption within a year of study enrollment;
* History of immunosuppression/immune deficiency disorders (including human immunodeficiency virus (HIV) infection or acquired immunodeficiency syndrome (AIDS) or use of immunosuppressive medications;
* Significant concurrent illness, such as uncontrolled diabetes (with a hemoglobin A1C of more than 8) (i.e., any disease state that in the opinion of the Investigator would interfere with the anesthesia, treatment, or healing process);
* Mentally incompetent, prisoner or evidence of active substance or alcohol abuse;
* Any condition which, in the Investigator's opinion, would make it unsafe (for the subject or study personnel) to treat the subject as part of this research study;
* Participation in another interventional study with potential exposure to an investigational drug within past 30 days;
* Pregnant females, due to possible discomfort with the procedure even though the procedure is localized and there is no new drug.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Estimated)
Dates: Start 2021-01-19 (Actual); Primary Completion 2028-03 (Estimated); Study Completion 2028-12 (Estimated)

PRIMARY OUTCOMES:
Change in the CTCAE (National Cancer Institute Common Terminology Criteria for Adverse Events v5) grading | 12 months
  Patients will receive a grading for their treated radiation wound based on the CTCAE. Changes in the grading over time will be used to assess improvement of the wound

CONTACTS AND LOCATIONS:
Overall Officials: Yen-Lin E Chen, MD, Principal Investigator — Massachusetts General Hospital
Locations (1):
- Massachusetts General Hospital, Wellman Center for Photomedicine, Boston, Massachusetts, United States